CLINICAL TRIAL: NCT00337402
Title: Effects of Gastrostomy on Quality of Life and Survival in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Effects of Gastrostomy on Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Angers (Other Government); University Hospital, Bordeaux (Other); University Hospital, Caen (Other); University Hospital, Grenoble (Other); University Hospital, Lille (Other); University Hospital, Limoges (Other); Neurological department of Lyon University Hospital (Unknown); University Hospital, Marseille (Other); University Hospital, Montpellier (Other); Central Hospital, Nancy, France (Other); Centre Hospitalier Universitaire de Nice (Other); University Hospital, Paris (Other); University Hospital, Strasbourg (Other); University Hospital, Toulouse (Other); University Hospital, Tours (Other)
Other Study IDs: CHU63-0001
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Gastrostomy; Quality of life
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Results about effects of symptomatic treatment on QoL appears conflicting in ALS patients. Moreover no clear effects of gastrotomy have be shown on survival. Prospective study on effect of tube feeding, QoL and survival is performed in 17 teaching hospitals in France (observational study)

DETAILED DESCRIPTION:
Following data have been recorded each three months: QoL (MOS-SF 36 and ALSAQ), bodily mass index, testing and ALS-FRS scale, functional respiratory measures, impedance analysis, and the time for tube feeding procedure, the conditions of the acceptance and side-effects of gastrotomy

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years-old
* ALS certain or probable
* vital capacity (respiratory) > 70 %
* under riluzole

Exclusion Criteria:

* ALS in family
* other conditions affected survival and QoL
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380
Dates: Start 2002-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Clavelou, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, France